CLINICAL TRIAL: NCT03191838
Title: Audiovisual Distraction Versus Propofol Sedation for Patients Undergoing Total Knee or Hip Replacement Surgery Under Spinal Anesthesia
Brief Title: Audiovisual Distraction for Patients Undergoing Total Knee or Hip Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102391
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audiovisual (Experimental): The interventional group will be given audiovisual equipment. An Apple iPad will be attached to a Mayo stand and placed approximately 12-15 inches from the patient's face. Noise canceling headphones will be connected to the iPad. A movie of the subject's choosing will be shown on the iPad with a comfortable level of sound.
  Interventions: Other: Audiovisual Distraction
- Controls (No Intervention): The control group will not be given distraction equipment.

INTERVENTIONS:
Other: Audiovisual Distraction — The interventional group will be given audiovisual equipment. An Apple iPad will be attached to a Mayo stand and placed approximately 12-15 inches from the patient's face. Noise canceling headphones will be connected to the iPad. A movie of the subject's choosing will be shown on the iPad with a comfortable level of sound.
  Arms: Audiovisual

SUMMARY:
The primary purpose of this study is to investigate whether audiovisual distraction can lead to a reduction in standard of care administered intraoperative propofol consumption compared to those who receive propofol sedation alone in adults having total hip or knee replacement surgery under spinal anesthesia.

DETAILED DESCRIPTION:
The perioperative period is often anxiety-provoking experience for many of our patients. Pain and awareness are the two primary concerns voiced most frequently. For total knee and hip replacement surgery, we offer our patients a spinal anesthetic which produces complete sensory blockade below the level of the waist. Despite a completely insensate knee or hip, patients still desire sedation during the surgery in order to remain unaware of their surgical surroundings. Propofol is commonly used in these monitored anesthesia care procedures because of its favorable drug profile. However, we have observed that anesthesia providers often use high infusion rates of propofol in order to achieve 'adequate patient comfort'. In this scenario, providers are often left with the dilemma of providing deeper levels of sedation for a pleasant patient experience and dealing with the potential cardiorespiratory complications that follow from oversedation. Unwanted side-effects include respiratory depression, airway obstruction and hypotension. Clinicians have began looking for other non-pharmacological ways to provide safe anxiolysis in the operating room while avoiding these undesirable side-effects.

Previous studies have shown that audiovisual distraction (AVD) can reduce stress and anxiety during the perioperative period. In 1997, Ganapathy et al. examined the use of sedative medications in elderly patients undergoing orthopedic procedures under spinal anesthesia. They compared patient-controlled propofol administration and anesthesiologist-controlled midazolam and fentanyl administration.This study found that there were no differences in patient satisfaction between the two groups. The secondary outcomes did show that propofol consumption was associated with significantly more episodes of brief respiratory rate depression but did not increase the need for emergency airway interventions.1

Ayoub et al studied propofol consumption in patients undergoing orthopedic procedures under spinal anesthesia using auditory distraction. This study demonstrated that auditory distraction decreased the amount of propofol consumed in patients using auditory distraction compared to those who had propofol sedation alone.2

Lee et al. began to shift the paradigm of medication induced anxiolysis and pain control during painful procedures through a series of studies examining different forms of distraction. An initial study conducted by this group confirmed that audio distraction during stimulating procedures (colonscopies) reduced the amount of propofol required. In 2003, they combined audio and visual distraction in patients undergoing and compared the dosages of propofol required to patients having only visual distraction or no distraction. This study found that patients with both audio and visual distraction required significantly less propofol than patients receiving visual distraction or patient-controlled sedation alone. Other key findings in the AVD group included reduced procedure time, a greater willingness by the patient to repeat the procedure under the same circumstances, and a statistically significant higher satisfaction score with the process.3

None of these studies has attempted to evaluate a possible reduction in propofol consumption for patients having a spinal anesthetic with both audio and visual distraction. We believe the next step to improving the perioperative experience for our patients is to incorporate AVD for patients having total knee and hip replacement surgery under a spinal anesthetic. Our hypothesis is that AVD will significantly reduce standard of care administered propofol consumption while still providing a pleasant experience for our patients and reducing unwanted side-effects associated with higher levels of propofol sedation.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years of age having a
* Primary total hip or knee arthroplasty
* Surgery under a spinal anesthetic

Exclusion Criteria:

* ASA status >3
* parturients
* documented hearing or vision loss
* chronic opioid use (>30mg PO MEQ daily for >1 month)
* diagnosis of OSA, contraindications to spinal (coagulopathy, infection, spinal hardware)
* non-English speaking
* current history of substance abuse
* schizophrenia
* generalized anxiety disorder
* Alzheimer's disease
* other dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Propofol Consumption | Intra-operative drug use
  Comparison of AV distraction patients and control group propofol consumption (micrograms/kilograms/minute) during surgery

SECONDARY OUTCOMES:
Movement | continuously monitored during surgery every fifteen minutes
  Graded movement during surgery using a validated movement scale graded 0-3 with 0 being no movement and 3 being surgery difficult to perform
Satisfaction with Anesthesia | Post-operatively obtained directly following admission to a phase II anesthesia care unit
  Iowa Satisfaction with Anesthesia score, a validated assessment of patient reported undesirable effects from surgery and if they would have the same anesthetic in future surgeries
provider-involved airway interventions | continuously monitored during surgery
  The number and timing of provider-involved airway interventions including replacement of nasal cannula with facemask, placement of oral or nasal airway, or endotracheal intubation will be recorded
hypotensive episodes | continuously monitored during surgery
  hypotensive episodes including SPB less than 90
oxygen desaturation episodes | continuously monitored during surgery
  oxygen desaturation episodes including SPO2 less than 90

CONTACTS AND LOCATIONS:
Overall Officials: Adam Meier, DO, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers